CLINICAL TRIAL: NCT07214155
Title: Effects of Various Cannabis Strains on Perceptual, Subjective and Objective Use Outcomes
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB00529431; R01DA059584 (NIH)
Record Dates: First submitted 2025-10-03; First posted 2025-10-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Cannabis Intoxication
Keywords: Cannabis; Indica; Sativa
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols; Dronabinol

STUDY DESIGN:
Intervention Model Description: All participants will complete all dose conditions (study arms) in a randomized order
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Indica-Labeled Cannabis - Placebo (Placebo Comparator): Participants administer smoked cannabis labeled as indica containing 0mg THC.
  Interventions: Drug: Cannabis; Other: 0 mg THC (placebo)
- Sativa-Labeled Cannabis - Placebo (Placebo Comparator): Participants administer smoked cannabis labeled as Sativa containing 0mg THC.
  Interventions: Drug: Cannabis; Other: 0 mg THC (placebo)
- Generically-Labeled Cannabis - Placebo (Placebo Comparator): Participants administer smoked cannabis labeled generically containing 0mg THC.
  Interventions: Drug: Cannabis; Other: 0 mg THC (placebo)
- Indica-Labeled Cannabis - Active (Experimental): Participants administer smoked cannabis labeled as indica containing 25mg THC.
  Interventions: Drug: Cannabis
- Sativa-Labeled Cannabis - Active (Experimental): Participants administer smoked cannabis labeled as sativa containing 25mg THC.
  Interventions: Drug: Cannabis
- Generically-Labeled Cannabis - Active (Experimental): Participants administer smoked cannabis labeled generically containing 25mg THC.
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis — Cannabis will be administered via smoked inhalation.
Other: 0 mg THC (placebo) — 0 mg THC (placebo)
  Arms: Generically-Labeled Cannabis - Placebo; Indica-Labeled Cannabis - Placebo; Sativa-Labeled Cannabis - Placebo

SUMMARY:
This study will evaluate the subjective and behavioral effects of cannabis products labeled as indica, sativa, or generic.

DETAILED DESCRIPTION:
This clinical laboratory study will be double-blind, placebo-controlled and will utilize a within-subjects experimental design. Participants will complete 6 outpatient drug administration sessions that will consist of self-administration of smoked cannabis (0, or 25mg THC) labeled as indica, sativa, or generically-labelled. Primary outcomes include performance on cognitive and psychomotor assessments, subjective drug effects, and simulated driving performance. Smoking topography will also be characterized.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent.
* Be between the ages of 21 and 55
* Be in good general health based on a physical examination, medical history, vital signs, and screening urine and blood tests
* Test negative for drugs of abuse including breath alcohol at the screening visit and at clinic admission
* Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at clinic admission. Participants must confirm use of appropriate birth control methods (e.g., condoms, birth control pills) throughout the entirety of the study.
* Blood pressure at Screening Visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg
* Have prior experience smoking cannabis but not currently using more than 3 times per week on average; participants must be active cannabis users (i.e., report past 3-month use) to participate.

Exclusion Criteria:

* Self-reported use of illicit drugs (e.g., amphetamine, cocaine, methamphetamine, 3,4-Methylenedioxymethamphetamine (MDMA), lysergic acid diethylamide (LSD), ketamine, heroin, psilocybin, prescription medications not prescribed to the person) in the past 30 days.
* History of or current evidence of significant medical (e.g., seizure disorder) or psychiatric illness (e.g. psychosis) judged by the investigator to put the participant at greater risk of experiencing an adverse event due to exposure or completion of other study procedures.
* History of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina).
* Enrolled in another clinical trial or having received any drug as part of a research study within 30 days prior to dosing.
* Having previously sought medical attention to manage adverse effects following acute cannabis use
* Individuals with anemia or who have donated blood in the prior 30 days

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Number of Correct Trials on Paced Auditory Serial Addition Task (PASAT) | Baseline, 0-, 1-, 1.5-, 2-, 3-, 4-, 5-, and 6-hours post-dosing
  Computerized version of Paced Auditory Serial Addition Task will be administered to assess working memory performance. Will report the total correct trials out of 90 recorded (lower scores indicate worse performance).
Driving Under the Influence of Drugs (DRUID) application global impairment score | Baseline, 0-, 1-, 1.5-, 2-, 3-, 4-, 5-, and 6-hours post-dosing
  Acute cognitive and behavioral impairment will be assessed with global impairment score(range 0-100) on the DRUID app (higher scores indicate greater impairment).
Number of Correct Trials on the Digit Symbol Substitution Task (DSST) | Baseline, 0-, 1-, 1.5-, 2-, 3-, 4-, 5-, and 6-hours post-dosing
  Computerized version of Digit Symbol Substitution Task will be administered to assess psychomotor performance. Will report the total correct trials in 90 seconds (lower scores indicate worse performance).
Biphasic alcohol effects scale (BAES) - Sedative Score | Baseline, 0-, 0.5-, 1-, 1.5-, 2-, 3-, 4-, 5-, and 6-hours post-dosing
  The BAES is used to assess sedative and stimulant subjective effects of alcohol. It has been shown to be sensitive to the effects of cannabis too. There are 7 sedative-related questionnaire items, each presented on a scale of 0 (not at all) to 10 (extremely), which are integrated to produce an overall sedative score (0-70). Higher score more effects.
Biphasic alcohol effects scale (BAES) - Stimulant Score | Baseline, 0-, 0.5-, 1-, 1.5-, 2-, 3-, 4-, 5-, and 6-hours post-dosing
  The BAES is used to assess sedative and stimulant subjective effects of alcohol. It has been shown to be sensitive to the effects of cannabis too. There are 7 stimulant-related questionnaire items, each presented on a scale of 0 (not at all) to 10 (extremely), which are integrated to produce an overall stimulant score (0-70). Higher score more effects.
Driving performance as assessed by standard deviation of lateral position (SDLP) | Baseline, 0-, 2-, 4-, and 6-hours post dosing.
  The STISIM Drive® M4000-R Console system will be used to assess driving performance, a state-of-the-art technology that has been independently validated to reflect real-world driving conditions. SDLP (measured in cm) will be determined during each drive. This measure is a composite index of lateral control and incorporates lane weaving, swerving, and over-correcting. SDLP is the gold standard of quantifying the magnitude of driving impairment from drugs and alcohol and has excellent predictive validity to actual driving. Scores range from 0 to no upper limit. Higher scores represent higher magnitude of driving impairment.
Driving performance as assessed by global drive score | Baseline, 0-, 2-, 4-, and 6-hours post dosing.
  Driving impairment will be assessed via a composite drive score (higher scores indicate greater impairment). The composite drive score is derived by integrating various driving outcomes (see primary and secondary driving outcomes). There is no upper or lower limit to possible scores
Drug Effect Questionnaire (DEQ) - Feel Drug Effect | Baseline, 0-, 0.5-, 1-, 1.5-, 2-, 3-, 4-, 5-, and 6-hours post-dosing
  The DEQ will be used to obtain subjective ratings of "feel drug effects". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effect Questionnaire - Confidence to Drive | Baseline, 0-, 0.5-, 1-, 1.5-, 2-, 3-, 4-, 5-, and 6-hours post-dosing
  The DEQ will be used to obtain subjective ratings of "confidence to drive". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effect Questionnaire - Alert | Baseline, 0-, 0.5-, 1-, 1.5-, 2-, 3-, 4-, 5-, and 6-hours post-dosing
  The DEQ will be used to obtain subjective ratings of "alert". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Drug Effect Questionnaire - Sleepy/Tired | Baseline, 0-, 0.5-, 1-, 1.5-, 2-, 3-, 4-, 5-, and 6-hours post-dosing
  The DEQ will be used to obtain subjective ratings of "sleepy/tired". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.

SECONDARY OUTCOMES:
Drug Effect Questionnaire - Like Drug Effect | Baseline, 0-, 0.5-, 1-, 1.5-, 2-, 3-, 4-, 5-, and 6-hours post-dosing
  The DEQ will be used to obtain subjective ratings of "like drug effect". Score range from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Anticipated Effects of Cannabis Scale (AECS) - Creative | Baseline prior to drug administration
  The AECS will be used to obtain subjective ratings of "creative". Score range from 0 (none) to 10 (extreme) using a 10mm line anchored with none/extreme designation.
Anticipated Effects of Cannabis Scale (AECS) - Drowsy | Baseline prior to drug administration
  The AECS will be used to obtain subjective ratings of "Drowsy". Score range from 0 (none) to 10 (extreme) using a 10mm line anchored with none/extreme designation.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zamarripa, PhD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No